CLINICAL TRIAL: NCT02886637
Title: Effects of Immune Function on Prognositic Outcome in Critical Ill Patients With Acinetobacter Baumannii Infection
Status: Completed | Type: Observational
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jianfeng Xie, Attending, Southeast University, China
Other Study IDs: 20160826
Record Dates: First submitted 2016-08-27; First posted 2016-09-01 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Acinetobacter Baumannii Infection
Keywords: A baumannii infection; Immunosuppression; prognosis; immune function

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acinetobacter baumannii infection: Critically ill patients infect with Acinetobacter baumannii
  Interventions: Other: None intervention

INTERVENTIONS:
Other: None intervention

SUMMARY:
The purpose of the present study is to evaluate the effects of immune function on prognositic outcome in critical ill patients with Acinetobacter baumannii infection.

DETAILED DESCRIPTION:
This is a single-center, observational study. Patients with Acinetobacter baumannii infection in the intensive care unit of Zhongda Hospital were enrolled. We recorded the data of age, ICU admission diagnosis, underlying diseases, APACHE II score and infection site. Body temperature, heart rate, white blood cell counts, procalcitonin, C-reactive protein, SOFA score and the level of CD4+, CD8+, Th1, Th2 and HLA-DR in the blood measured by flow cytometry on the D1, D3 and D7 were also recorded.We can get the results of the change of immune function of critical ill patients after Acinetobacter baumannii infection. After compare the patients who die of survive at 28 day after infection, we can get the results of the relationship between the immune function and the outcome. We also can calculate the effect immune function on prognositic mortality in patients with Acinetobacter baumannii infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to ICU
* Infection with Acinetobacter baumannii
* Agree to participate the study

Exclusion Criteria:

* Age less than 16 years old or older than 80 years old
* pregnancy
* immunosuppression patients which include

  1. therapy 0.5mg/kg/day of prednisoneover(equivalent dose of other glucocorticoids) for at least 1 month within recent 3 month
  2. Cancer chemotherapy within recent 3 month
  3. Receive immunosuppression treatment because of solid organ transplant or Autoimmune diseases
  4. allogeneic bone marrow transplantation or allogeneic haematopoietic stem cell transplantation.
  5. HIV infection

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who admitted into ICU and infection with Acinetobacter baumannii.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
28 day mortality | 28 day

IPD SHARING:
Plan to Share IPD: Yes
we would like to share our data. Someone who need data can contact us with Email.